CLINICAL TRIAL: NCT04896853
Title: Treatment of Respiratory Complications Associated With COVID-19, Influenza A, Metapneumovirus, Respiratory Syncytial Virus Infection Using Wharton's Jelly-Umbilical Cord Mesenchymal Stromal Cells (ProTrans®): Open Phase IB Clinical Trial
Brief Title: Treatment of Respiratory Complications Associated With COVID19,Influenza ,Metapneumovirus,RSV Infection Using ProTrans®
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NextCell Pharma Ab (Industry)
Collaborators: Karolinska Trial Alliance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO TRANS 19+; 2020-002078-29 (EudraCT Number)
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Influenza A; Metapneumovirus Pneumonia; Respiratory Syncytial Virus (RSV)

STUDY DESIGN:
Intervention Model Description: This is an open, dose escalating Phase IB Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Wharton's Jelly (WJ)-Umbilical Cord (UC) Mesenchymal Stromal Cells (ProTrans®).Study patients 1-3 will receive a single dose of 25 million cells, patients 4-6 will receive 100 million cells and patients 7-9 will receive 200 million cells.
  Interventions: Biological: ProTrans®

INTERVENTIONS:
Biological: ProTrans® — Allogeneic Wharton's jelly (WJ) Mesenchymal Stromal Cells

SUMMARY:
To investigate the safety and tolerance of a single infusion of ProTrans® in subjects with "severe" respiratory complications associated with pneumonia caused by COVID-19, Influenza A, Metapneumovirus or RSV infection.

DETAILED DESCRIPTION:
The investigators hypothesize that the systemic delivery of WJ-MSCs exerts an anti-inflammatory action and anti-apoptotic effect in the lung of COVID-19, Influenza A, Metapneumovirus or RSV patients. The nature of these cells to immunomodulate both tissue resident and bloodborne immune cells towards a more anti-inflammatory and tolerogenic profile, results in a reduction of tissue-based inflammation within the lung and triggering of repair responses. This clinically culminates in a beneficial action on patients with "severe" respiratory complications associated with pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥18 years old
* Has laboratory-confirmed SARS-CoV-2, Influenza A, Metapneumovirus or RSV infection as determined by reverse-transcription polymerase chain reaction (RT-PCR) in any specimen prior to inclusion.
* Hospitalized patients.
* Patients classified as severe pneumonia, as defined by the need for continuous supplemental oxygen 5 L/min 02 OR high flow oxygen, 35% FiO2 > 30l/min and cannot saturate > 96% NOT under "non-invasive" ventilation NOR invasive mechanical ventilation NOR ECMO.
* Women of childbearing potential must agree to use contraception or acceptable birth control for the duration of the study. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation 1:

  * oral
  * intravaginal
  * transdermal, progestogen-only hormonal contraception associated with inhibition of ovulation 1:
  * oral
  * injectable
  * implantable 2; intrauterine device (IUD) 2, intrauterine hormone-releasing system (IUS) 2, bilateral tubal occlusion 2, vasectomised partner 2,3, sexual abstinence 4

    1. Hormonal contraception may be susceptible to interaction with the Investigational Medicinal Products (IMP), which may reduce the efficacy of the contraception method
    2. Contraception methods that in the context of this guidance are considered to have low user dependency.
    3. Vasectomised partner is a highly effective birth control method provided that partner is the sole sexual partner of the trial participant and that the vasectomised partner has received medical assessment of the surgical success. 4 In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
* Provision of a written informed consent

Exclusion Criteria:

* Inability to provide informed consent
* Patients not expected to survive for 24 hours or mechanically ventilated at inclusion or previously during present hospitalization
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotrophin (hCG) laboratory test
* Patients with BMI ≥30
* Patients with known, or previous, malignancy
* Patients with other serious systemic diseases deemed of contra-indication by the physician
* Patient with any of following laboratory results out of the ranges detailed below at screening: Absolute neutrophil count (ANC) ≤ 1.0 x 10e9/L, Platelets (PLT) < 50 10e9 /L, ASAT or ALAT > 5N, estimated glomerular filtration rate (eGFR) < 30 mL/min
* Current documented bacterial infection
* Serological evidence of infection with human immunodeficiency virus, Treponema pallidum, hepatitis B antigen (serology consistent with previous vaccination and a history of vaccination is acceptable) or hepatitis C
* Latent or previous as well as on-going therapy against tuberculosis, or exposed to tuberculosis or have travelled in areas with high risk of tuberculosis or mycosis within the last 3 months
* Patients with known allergies to a component of the ProTrans® product
* Ongoing treatment with Remdesivir
* Pre-existing chronic respiratory diseases requiring long- term oxygen therapy
* Pre-existing cirrhosis with basal Child and Pugh of C
* Patients with history of increased risk for thrombo- embolic and/or co-morbidity for thrombo- embolism
* Patients with a history of myocardium infarction
* A history of cardiac dysfunction, as assessed as:

Clinical sign of a congestive heart failure refractory; Left ventricular ejection fraction <35% at myocardial scintigraphy or echocardiography; Pulmonary arterial hypertension with systolic pulmonary artery pressure (PAP) at echography > 40 mmHg Chronic atrial fibrillation requiring oral anticoagulant therapy; Uncontrolled ventricular arrhythmia; Pericardial effusion with hemodynamic compromise assessed by echocardiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerance of a single infusion of ProTrans® | 24 months
  Grade 3 or 4 adverse event but not usual in natural course of the disease.

SECONDARY OUTCOMES:
Effect of ProTrans® -MSC on patient clinical status, including mortality, at day 7 | 7 days
  Effect of ProTrans® -MSC on patient clinical status as assessed on the 7-point ordinal scale; 1. Not hospitalized, no limitations on activities 2. Not hospitalized, limitation on activities 3. Hospitalized, not requiring supplemental oxygen 4. Hospitalized, requiring supplemental oxygen 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices 6. Hospitalized, on invasive mechanical ventilation or Extracorporeal membrane oxygenation (ECMO) 7. Death.
Effect of ProTrans® -MSC on patient clinical status, including mortality, at day 15 | 15 days
  Effect of ProTrans® -MSC on patient clinical status as assessed on the 7-point ordinal scale; 1. Not hospitalized, no limitations on activities 2. Not hospitalized, limitation on activities 3. Hospitalized, not requiring supplemental oxygen 4. Hospitalized, requiring supplemental oxygen 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices 6. Hospitalized, on invasive mechanical ventilation or ECMO 7. Death.
Effect of ProTrans® -MSC on patient clinical status, including mortality, at day 30 | 30 days
  Effect of ProTrans® -MSC on patient clinical status as assessed on the 7-point ordinal scale; 1. Not hospitalized, no limitations on activities 2. Not hospitalized, limitation on activities 3. Hospitalized, not requiring supplemental oxygen 4. Hospitalized, requiring supplemental oxygen 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices 6. Hospitalized, on invasive mechanical ventilation or ECMO 7. Death.
Time to clinical improvement after ProTrans® - MSC infusion | 30 days
  Time to clinical improvement of one category from admission on the 7-point ordinal scale after ProTrans® - MSC infusion
Effect of of ProTrans® -MSC on lung damage | Up to 60 days
  Lung damage examination using imaging techniques (Chest X ray/CT scan /or on doppler ultrasound) when assessed for clinical need up to hospital discharge X ray/CT scan /or on doppler ultrasound) when assessed for clinical need
Duration of hospitalization and Intensive Care Unit (ICU) stay | Up to 60 days
  Duration of hospitalization and ICU stay
Kinetics of COVID-19, Influenza A, Metapneumovirus, Respiratory Syncytial Virus (RSV) viral load after ProTrans® -MSC infusion | Up to 30 days
  Quantitative PCR for SARS-CoV, Influenza A, Metapneumovirus, Respiratory Syncytial Virus (RSV) virus in throat swabs (time frame: before MSC infusion on Day 0 and after MSC infusion on day 30)
Evolution of biological markers of liver, myocardium and inflammation | Up to 24 months
  Evaluation of different biomarker after ProTrans® -MSC infusion
Tolerance of allogeneic Wharton's jelly (WJ) Mesenchymal Stromal Cells (ProTrans®) for severe COVID-19, Influenza A, Metapneumovirus or RSV respiratory conditions | Up to 24 months
  Investigation of tolerance of Wharton's jelly (WJ) Mesenchymal Stromal Cells (ProTrans®) for treatment of viral respiratory tract infections

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Svahn, PhD, Study Chair — NextCell Pharma; Josefine Sundh, MD, Principal Investigator — Department of Cardiology, Respiratory medicine and Physiology, Örebro University Hospital
Locations (1):
- Department of Cardiology, Respiratory medicine and Physiology, Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No